CLINICAL TRIAL: NCT00100698
Title: Physiologic Growth Hormone Effects in HIV Lipodystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Steven Grinspoon, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DK63639; R01DK063639 (NIH)
Record Dates: First submitted 2005-01-04; First posted 2005-01-05 (Estimated); Results first posted 2010-07-22 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: AIDS; HIV Infections
Keywords: HIV; lipodystrophy; growth hormone; visceral fat; IGF-I; Treatment Experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Lipodystrophy | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): recombinant human growth hormone subcutaneously once a day
  Interventions: Drug: recombinant human growth hormone
- 2 (Placebo Comparator): placebo subcutaneously once a day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: recombinant human growth hormone — growth hormone dosed by weight and IGF-1 level,subcutaneously once a day, 18 months
  Other Names: Serostim
  Arms: 1
Drug: placebo — placebo subcutaneously once a day, 18 months
  Arms: 2

SUMMARY:
This study will investigate long-term, low-dose growth hormone administration in HIV-infected patients with reduced growth hormone (GH) secretion and increased visceral adiposity. We hypothesize that low-dose growth hormone will reduce visceral fat. Secondary endpoints will include measures of insulin-like growth factor-1 (IGF-1), glucose homeostasis, lipids, blood pressure,bone density, cardiovascular risk and safety parameters.

DETAILED DESCRIPTION:
This study will investigate long-term, low-dose growth hormone administration in HIV-infected patients with reduced growth hormone (GH) secretion and increased visceral adiposity. We hypothesize that low-dose growth hormone will reduce visceral fat preferentially over subcutaneous fat, and increase lean body mass. Secondary endpoints will include measures of IGF-1, glucose homeostasis, lipids, blood pressure,bone density, cardiovascular risk and safety parameters. Dosing of growth hormone will be based on patients' IGF-1 levels and will not exceed 6mcg/kg/day.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18-60
* Previously diagnosed HIV infection
* Stable antiviral regimen for at least 12 weeks prior to enrollment
* Waist-to-hip ratio >0.90 for men and >0.85 for women
* Evidence of at least one of the following recent changes: *increased abdominal girth,

  *relative loss of fat in the extremities, *relative loss of fat in the face
* Simulated peak GH response to arginine/GHRH of less than 7.5 mcg/dL

Exclusion Criteria:

* Use of Megace, anti-diabetic agents, GH, or other anabolic agents, pharmacologic glucocorticoid (prednisone >5 mg/day or its equivalent) for 3 months prior to enrollment. Patients on a standard dose of testosterone for documented hypogonadism will be allowed to enter the protocol. Women taking standard estrogen replacement therapy for >3 months will be allowed in the study.
* Diabetes mellitus
* Other severe chronic illness
* HgB <9.0 g/dL, creatinine >1.4 mg/dL, or PSA >4 ng/mL
* Positive BHCG or failure to use appropriate birth control during study. Acceptable methods include oral contraceptives, depo provera or combined progesterone-estrogen injections, transdermal contraceptive patches, IUD's, barrier devices (condoms, diaphragms), and abstinence.
* Carpal tunnel syndrome
* Active malignancy or history of pituitary malignancy, history of colon cancer or prostate malignancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2004-01; Primary Completion 2007-10 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grinspoon, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Lo J, You SM, Canavan B, Liebau J, Beltrani G, Koutkia P, Hemphill L, Lee H, Grinspoon S. Low-dose physiological growth hormone in patients with HIV and abdominal fat accumulation: a randomized controlled trial. JAMA. 2008 Aug 6;300(5):509-19. doi: 10.1001/jama.300.5.509. PMID 18677023

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with HIV and lipodystrophy were recruited between November 2003 and March 2006 via community advertisement, HIV support and advocacy groups, and infectious disease or primary care physician referral.
Pre-assignment Details: Patients who do not meet growth hormone inclusion criteria were excluded from the trial before assignment to groups.
Groups:
- Recombinant Human Growth Hormone: recombinant human growth hormone starting at 2 micrograms/kilograms/day subcutaneously and increased to maximum dose of 6 micrograms/kilograms/day subcutaneously
- Placebo: placebo subcutaneously once a day
Period: Overall Study
Arm/Group | Recombinant Human Growth Hormone | Placebo
Started | 27 | 29
Completed | 21 | 27
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recombinant Human Growth Hormone | Placebo | Total
Number analyzed (Participants) | 27 | 29 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 29 | 56
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 46.7 (7.9) | 47.4 (6.1) | 47.1 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 26 | 26 | 52
Region of Enrollment [Number; unit: participants]
  United States | 27 | 29 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change in Visceral Adipose Tissue Area From Baseline to 18 Months
Description: change in visceral adipose tissue area as measured by single-slice abdominal computed tomographic scan
Time Frame: 18 months
Measure: Mean (Standard Error); unit: centimeters squared
Arm/Group | Recombinant Human Growth Hormone | Placebo
Number analyzed (Participants) | 27 | 29
centimeters squared | -22 (6) | -4 (4)
Statistical Analysis 1: Comparison: Recombinant Human Growth Hormone vs Placebo; Test type: Superiority or Other; p = 0.049, repeated measures mixed effects ANCOVA; Mean Difference (Net) = -22, 95% CI 2-sided [-38 to -0.5], Standard Error of Mean 6

2. Secondary Outcome: Change in Insulin-like Growth Factor-I From Baseline to 18 Months
Description: Change in insulin-like growth factor-1
Time Frame: 18 months
Measure: Mean (Standard Error); unit: nanograms/milliliter
Arm/Group | Recombinant Human Growth Hormone | Placebo
Number analyzed (Participants) | 27 | 29
nanograms/milliliter | 109 (11) | -25 (8)

3. Secondary Outcome: Change in Trunk Fat
Time Frame: 18 months
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Recombinant Human Growth Hormone | Placebo
Number analyzed (Participants) | 27 | 29
kilograms | -0.5 (0.2) | 0.2 (0.2)

4. Secondary Outcome: Change in Fasting Glucose
Description: change in fasting glucose
Time Frame: 18 months
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Recombinant Human Growth Hormone | Placebo
Number analyzed (Participants) | 27 | 29
mg/dL | 6 (1) | 5 (1)

5. Secondary Outcome: Change in Trunk to Extremity Ratio
Description: change in trunk to extremity ratio
Time Frame: 18 months
Measure: Mean (Standard Error); unit: kilogram per kilogram
Arm/Group | Recombinant Human Growth Hormone | Placebo
Number analyzed (Participants) | 27 | 29
kilogram per kilogram | -0.4 (0.1) | 0 (0)

6. Secondary Outcome: Change in Triglycerides
Description: Change in triglycerides
Time Frame: 18 months
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Recombinant Human Growth Hormone | Placebo
Number analyzed (Participants) | 27 | 29
mg/dL | -7 [-43 to 41] | 0 [-56 to 51]

7. Secondary Outcome: Change in Subcutaneous Adipose Tissue
Description: Change in subcutaneous adipose tissue
Time Frame: 18 months
Measure: Mean (Standard Error); unit: centimeters squared
Arm/Group | Recombinant Human Growth Hormone | Placebo
Number analyzed (Participants) | 27 | 29
centimeters squared | 4 (4) | 4 (4)

8. Secondary Outcome: Change in CD4 Cells
Description: Change in CD4 cells
Time Frame: 18 months
Measure: Mean (Standard Error); unit: cells/microliter
Arm/Group | Recombinant Human Growth Hormone | Placebo
Number analyzed (Participants) | 27 | 29
cells/microliter | -19 (13) | 15 (21)

9. Secondary Outcome: Change in Logarithm HIV Viral Load
Description: Change in logarithm base 10 HIV viral load
Time Frame: 18 months
Measure: Mean (Standard Error); unit: log base 10 copies of RNA/milliliter
Arm/Group | Recombinant Human Growth Hormone | Placebo
Number analyzed (Participants) | 27 | 29
log base 10 copies of RNA/milliliter | 0 (0.1) | 0 (0.2)

10. Secondary Outcome: Change in Lean Body Mass
Description: change in lean body mass
Time Frame: 18 months
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Recombinant Human Growth Hormone | Placebo
Number analyzed (Participants) | 27 | 29
kilograms | 0.8 (0.3) | -0.5 (0.3)

11. Secondary Outcome: Change in Quality of Life Score From the Medical Outcomes Study-HIV Survey From Baseline to 18 Months
Description: Change in quality of life score was measured by the Medical Outcomes Study-HIV (MOS-HIV)survey. The MOS-HIV asks patients to report on health-related quality of life and physical function from the past 4 days. The scoring range is 0-100, and a higher score indicates better quality of life.
Time Frame: 18 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Recombinant Human Growth Hormone | Placebo
Number analyzed (Participants) | 27 | 29
units on a scale | -4 (3) | -4 (3)

12. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change in diastolic blood pressure
Time Frame: 18 months
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Recombinant Human Growth Hormone | Placebo
Number analyzed (Participants) | 27 | 29
mm Hg | -3 (1) | 4 (1)

13. Secondary Outcome: Change in Adiponectin
Description: Change in adiponectin
Time Frame: 18 months
Measure: Mean (Standard Error); unit: mcg/mL
Arm/Group | Recombinant Human Growth Hormone | Placebo
Number analyzed (Participants) | 27 | 29
mcg/mL | 1.0 (0.3) | 0.5 (0.1)

14. Secondary Outcome: Change in Carotid Intima Media Thickness (IMT)
Description: change in carotid intima media thickness (IMT)
Time Frame: 18 months
Measure: Mean (Standard Error); unit: millimeter
Arm/Group | Recombinant Human Growth Hormone | Placebo
Number analyzed (Participants) | 27 | 29
millimeter | 0.003 (0.008) | -0.003 (0.009)

15. Secondary Outcome: Change in Body Mass Index
Description: Change in body mass index
Time Frame: 18 months
Measure: Mean (Standard Error); unit: kilogram/meters squared
Arm/Group | Recombinant Human Growth Hormone | Placebo
Number analyzed (Participants) | 27 | 29
kilogram/meters squared | 0.2 (0.2) | 0.1 (0.1)

16. Secondary Outcome: Change in Extremity Fat
Description: Change in extremity fat
Time Frame: 18 months
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Recombinant Human Growth Hormone | Placebo
Number analyzed (Participants) | 27 | 29
kilograms | 0.3 (0.1) | 0.3 (0.1)

17. Secondary Outcome: Change in 2-hour Glucose
Description: Change in 2-hour glucose
Time Frame: 18 months
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Recombinant Human Growth Hormone | Placebo
Number analyzed (Participants) | 27 | 29
mg/dL | 16 (5) | -4 (4)

18. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic blood pressure
Time Frame: 18 months
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Recombinant Human Growth Hormone | Placebo
Number analyzed (Participants) | 27 | 29
mm Hg | -5 (2) | 1 (2)

ADVERSE EVENTS:
Time Frame: 18 months
Description: 1 participant in the growth hormone group dropped out of the study before ever receiving study drug and therefore was not included in the adverse event safety analysis.
Arm/Group | Recombinant Human Growth Hormone | Placebo
Serious Adverse Events (participants affected / at risk) | 4/26 | 1/29
Other Adverse Events (participants affected / at risk) | 3/26 | 5/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Human Growth Hormone (N=26) | Placebo (N=29)
rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
hospitalization (Infections and infestations) | 1 (1) | 0 (0) — hospitalization for confusion and transaminitis thought to be related to HIV disease progression
hip fracture requiring surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — hip fracture requiring surgery
appendicitis requiring surgery (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Human Growth Hormone (N=26) | Placebo (N=29)
tingling and paresthesia (Nervous system disorders) | 3 (3) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
hyperglycemia (Endocrine disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No